CLINICAL TRIAL: NCT07270835
Title: The Study of Zanubrutinib Combined With Rituximab in the Treatment of Secondary Hemophagocytic Lymphohistiocytosis in B-cell Lymphoma
Brief Title: Zanubrutinib Combined With Rituximab in the Treatment of Secondary HLH in B-cell Lymphoma
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Xuefeng He, professor, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HLH-003
Record Dates: First submitted 2025-11-18; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Hemophagocytic Lymphohistiocytosis; B Cell Lymphoma
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic; Lymphoma, B-Cell | interventions — Rituximab; zanubrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intervention group (Experimental): Rituximab 375 mg/m², intravenously, once weekly for 4 weeks (may be extended or adjusted according to clinical response).
  Zanubrutinib: 160 mg, orally, twice daily for 4 weeks as for rutuximab. Dose can be adjusted or extended according to tolerance and efficacy.
  When ≥3 grade hematological or intolerable non-hematological toxicity occur, zanubrutinib or rituximab will be suspended, and the dose will be reduced or resumed according to the toxicity grade after recovery. The dose of zanubrutinib should be adjusted according to the manufacturer's label with concomitant use of strong CYP3A inhibitor/inducer.
  Combined drugs: prednisone 100 mg/m²/d, orally, d1-5; Ruxolitinib 15mg bid orally; With/without emapalumab as appropriate.
  Interventions: Drug: Rituximab; Drug: Zanubrutinib

INTERVENTIONS:
Drug: Rituximab — 375 mg/m², intravenously, once weekly for 4 weeks
  Other Names: HALPRYZA
Drug: Zanubrutinib — 160 mg, orally, twice daily for 4 weeks as for rutuximab.
  Other Names: Brukinsa

SUMMARY:
For patients who met the inclusion criteria, treatment regimens were administered: Rituximab 375 mg/m², intravenously, once weekly for 4 weeks.

Zanubrutinib 160 mg, orally, twice daily for 4 weeks. Combined drugs: prednisone 100 mg/m²/d, orally, d1-5; Ruxolitinib 15mg bid orally; With/without emapalumab as appropriate.

DETAILED DESCRIPTION:
For patients who met the inclusion criteria, treatment regimens were administered:

Rituximab 375 mg/m², intravenously, once weekly for 4 weeks (may be extended or adjusted according to clinical response).

Zanubrutinib: 160 mg, orally, twice daily for 4 weeks as for rutuximab. Dose can be adjusted or extended according to tolerance and efficacy.

When ≥3 grade hematological or intolerable non-hematological toxicity occur, zanubrutinib or rituximab will be suspended, and the dose will be reduced or resumed according to the toxicity grade after recovery. The dose of zanubrutinib should be adjusted according to the manufacturer's label with concomitant use of strong CYP3A inhibitor/inducer.

Combined drugs: prednisone 100 mg/m²/d, orally, d1-5; Ruxolitinib 15mg bid orally; With/without emapalumab as appropriate.

ELIGIBILITY:
Inclusion Criteria:

* According to the diagnostic criteria of HLH-04, the patients meet the diagnostic criteria of HLH;
* HLH patients with definite or highly suspected evidence of B-cell lymphoma; Or HLH patients whose bone marrow flow cytometry show an increased proportion of CD20-positive B cells;
* Age of 14-80 years old, both sexes;
* Predicted survival beyond 1 month;
* Baseline serum creatinine ≤1.5 times ULN; Fibrinogen could be corrected to ≥0.6g/L by infusion;
* Negative serum HIV antibody; Either negative for HCV antibodies or positive for HCV antibodies but negative for HCV RNA. HBV surface antigen and HBV core antibody were negative. If any of the above was positive, HBV DNA titer in peripheral blood should be tested, and the titer was less than 1×10^3 copies /ml;
* Left ventricular ejection fraction (LVEF) ≥50% measured by echocardiography;
* The patient have no serious and uncontrollable infections, such as pulmonary infection, intestinal infection, and sepsis;
* Women of childbearing age must be confirmed to be not pregnant by pregnancy test and willing to take effective measures to prevent pregnancy during the study period and ≥12 months after the last dose; Pregnant and lactating women cannot participate; All male subjects took contraceptive measures during the trial and ≥3 months after the last dose;
* Patients should be able to sign informed consent.

Exclusion Criteria:

* Patients with known severe allergy to rituximab, zanubrutinib, or other BTK inhibitors;
* Severe active infections (including bacterial, viral or fungal infections) or uncontrolled co-infections;
* Severe organ dysfunction including NYHA class III-IV heart failure or severe arrhythmia; Liver function: ALT or AST >5 times the upper limit, or severe cirrhosis; Renal function: CrCl <30 mL/min or severe renal insufficiency;
* Combined with other malignant tumors and the expected survival time was less than 3 months;
* Have received other experimental drugs and had not completed the drug washout period;
* Pregnant or lactating women, or unwilling to use effective contraception;
* any condition that would not be suitable for participation in the study or that might affect adherence, follow-up, or safety assessment, as judged by the investigator.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
response rate of HLH after 4 weeks of treatment | after 4 weeks
  RR will be evaluated according to the response evaluation criteria recommended by the International Histiocyte Society.
OS at week 8 | after 8 weeks
  overall survival after 8 weeks of treatment

SECONDARY OUTCOMES:
AE | till the end of 4 weeks
  Adverse events will be evaluated according to NCI-CTCAE 5.0.
OS | at 4/8/12/24 weeks
  OS at 1/2/3 months/ 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Xuefeng He, doctor, Principal Investigator — department of hematology, The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided